CLINICAL TRIAL: NCT03274765
Title: Improved Medically Assisted Procreation (MAP) Monitoring
Brief Title: Improved Medically Assisted Procreation Monitoring
Acronym: NGAMP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC15_3019
Record Dates: First submitted 2017-08-31; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Infertility
Keywords: ovarian stimulation; blood test; Medically Assisted Procreation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with ovarian stimulation: Women followed in the MAP center of the Rennes University Hospital for ovarian stimulation monitoring Dosage of oestradiol
  Interventions: Diagnostic Test: Dosage of oestradiol

INTERVENTIONS:
Diagnostic Test: Dosage of oestradiol — The study is based on a concept using capillary blood tests using lateral flow by migration on membrane similarly to a pregnancy test, patented by a french company (NGBiotech).
  This study is therefore a feasibility study of a rapid test for oestradiol dosage during monitoring of ovarian stimulation.

SUMMARY:
Patient care in Medically Assisted Procreation (MAP) requires a close and regular monitoring of the evolution of the estradiol rate. This monitoring allows the dose and duration of treatment to be accurately adjusted for each woman (every 24 or 48 hours) up to 10 to 15 days of treatment with gonadotrophins. Oestradiol (E2) is secreted by the growing ovarian follicles and reflects their growth and maturity. Its plasma dosage makes it possible to monitor the ovarian response to stimulation.

This monitoring involves several constraints amongst which disruption of work life, stress, fatigue that can alter the response to treatment

DETAILED DESCRIPTION:
In order to improve the comfort of patients already under severe stress, simplification of this monitoring is proposed. The development of an immediate-release whole blood test for simplified monitoring of estradiol levels will provide considerable comfort in the management of patients. These patients are subjected to significant emotional and physical stress and the development of this test will reduce the negative consequences that result.

ELIGIBILITY:
Inclusion criteria:

* Women over 18 years old
* Patient followed for monitoring of ovarian stimulation;
* Having received information on the protocol and given consent to participate

Exclusion Criteria:

* Adult under safeguard of justice, guardianship or curatorship
* Persons deprived of liberty.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women followed in the MAP center of the Rennes University Hospital for ovarian stimulation monitoring
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-11-15 (Estimated); Primary Completion 2018-06-15 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
Rate of successful tests | 1 hour
  Number of tests yieling a result (whatever the value)

SECONDARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 month
  Rate of true positive test results (comparison with oestradiol level in blood sample, as gold standard)
Specificity | Through study completion, an average of 1 month
  Rate of true negative test results (comparison with oestradiol level in blood sample, as gold standard)

CONTACTS AND LOCATIONS:
Overall Officials: Celia RAVEL, MD, PhD, Study Director — CHU Rennes
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No